CLINICAL TRIAL: NCT04882475
Title: Biological Insights of First Relapsed-refractory Patients With Mantle Cell Lymphoma: the MANTLE-FIRST BIO Study.
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_MANTLE-FIRST BIO
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL (Mantle Cell Lymphoma); first relapsed-refractory patients; Histopathological characterization; Flow cytometry; NGS (Next Generation Sequencing); Gene Expression Profiling; RNA; BTKi (Bruton Tyrosine kinase inhibitors); Retrospective observational study; DNA
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For the primary objective of the study: Formaline-fixed paraffin-embedded (FFPE) material.
  For the secondary objectives of the study: viable cell suspensions, DNA extracted from Formaline-fixed paraffin-embedded (FFPE) tissue sections or frozen pellets, frozen cell suspensions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MCL patients relapsed or refractory to rituximab and induction chemotherapy with curative intent: An historical cohort of patients will be identified and selected both on a clinical base and according to the availability of Formaline-fixed paraffin-embedded (FFPE) material, frozen material or viable cryopreserved cells at Mantle Cell Lymphoma (MCL) diagnosis. Samples will be analyzed in 4 subgroups, each with different clinical specificity:
  1. refractory to Induction Chemoimmunotherapy (CIT);
  2. refractory to Bruton Tyrosine kinase (BTK) inhibitors (BTKi);
  3. sensitive to Induction Chemoimmunotherapy (CIT);
  4. sensitive to Bruton Tyrosine kinase (BTK) inhibitors (BTKi).

SUMMARY:
Retrospective observational study with a prospective biological evaluation of an historical cohort of first relapsed-refractory patients with mantle cell lymphoma who were relapsed or refractory to rituximab and chemotherapy containing induction regimens with curative intent.

DETAILED DESCRIPTION:
Biological samples from 80 Mantle Cell Lymphoma (MCL) patients will be collected and analyzed in 30 Italian sites in 36 months.

Patients will be identified and selected both on a clinical base and according to the availability of Formaline-fixed paraffin-embedded (FFPE) material, frozen material or viable cryopreserved cells at Mantle Cell Lymphoma (MCL) diagnosis. They will be analyzed in 4 subgroups, each with different clinical specificity: 1) refractory to Induction Chemoimmunotherapy (CIT); 2) refractory to Bruton Tyrosine kinase (BTK) inhibitors (BTKi); 3) sensitive to induction Induction Chemoimmunotherapy (CIT); 4) sensitive to BTK inhibitors (BTKi).

Each group will undergo central pathology revision with other immunohistochemical studies (Verona, Dr. Parisi; Milano, Prof. Ponzoni; Vicenza, Dr. D'Amore; Brescia, Prof. Facchetti). Formaline-fixed paraffin-embedded (FFPE) diagnostic specimens of Mantle Cell Lymphoma (MCL) will be screened by immunohistochemistry for the expression of immunoglobulin (Ig) heavy chains to identify Mantle Cell Lymphoma (MCL) cases lacking Immunoglobulin (Ig) expression.

Cytofluorimetric and molecular studies will be performed in the laboratories of the Verona University and at IFOM (Istituto FIRC di Oncologia Molecolare (FIRC = Fondazione Italiana per la Ricerca sul Cancro)). Specific methods will be used: Flow cytometry for the status of surface Ig expression and multiplexed phospho-specific flow cytometry, NGS (Next Generation Sequencing), Immunoglobulin (IgH/IgL V(D)J) profiling by BIOMED2 protocol-based, NGS (Next Generation Sequencing) technology in the relapsed-refractory mantle cell lymphoma (R/R MCL) cases, Chromatin accessibility studies by Assay for Transposase-Accessible Chromatin sequencing (ATAC-seq) (on viable cell suspensions or frozen pellets) and Gene Expression Profiling (GEP) by RNA-sequencing and RNA studies of the MALT1-MYC ((Mucosa-associated lymphoid tissue lymphoma translocation protein 1 - MYC) pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented diagnosis of Mantle Cell Lymphoma (MCL) as defined in the 2016 edition of the World Health Organization (WHO) classification, with available tissue for revision and additional studies;
* Diagnosis of Mantle Cell Lymphoma (MCL) between 1st of January 2008 and 30th of June 2020;
* Adults, 18-80 years at diagnosis;
* Relapsed or refractory disease after rituximab and chemotherapy containing induction regimens with curative intent.
* Treatment at relapse or progression on an intention-to-treat basis (ITT): at least one cycle of Chemo-immunotherapy (CIT), Bruton Tyrosine kinase inhibitors (BTKi), or alternative drugs combination;
* Subject understanding and voluntarily signing an informed consent form approved by an Independent Ethics Committee (IEC), prior to the initiation of any study-specific procedures.

Exclusion Criteria:

* Unavailability of the samples requested by the study;
* Any histology other than Mantle Cell Lymphoma (MCL);
* Patients treated with front line regimens containing only rituximab or with palliative therapy;
* Untreated patients; patients undergoing watchful waiting approach.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Mantle Cell Lymphoma (MCL) who were relapsed or refractory to rituximab and chemotherapy containing induction regimens with curative intent.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Histopathological characterization of patients with Mantle Cell Lymphoma (MCL) | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Histopathological characterization of patients with mantle cell lymphoma (MCL) who were relapsed or refractory to rituximab and chemotherapy containing induction regimens with curative intent. 80 Mantel Cell Lymphoma (MCL) patients stratified according to Chemo-immunotherapy (CIT) or Bruton Tyrosine kinase inhibitors (BTKi) resistance (20 for each of the groups previously identified) will undergo central pathology revision with assessment of Immunoglobulin (Ig) expression and other histopathological studies.

SECONDARY OUTCOMES:
Mutational analysis of Mantle Cell Lymphoma (MCL) driver genes | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Performed on formalin-fixed paraffin-embedded (FFPE) tissue sections as well as, when available, on frozen material or viable cryopreserved cells at Mantle Cell Lymphoma (MCL) diagnosis. The aim is to perform a mutational analysis for Mantle Cell Lymphoma (MCL) driver genes: Next Generation Sequencing (NGS) on approximately 80 cases of Mantle Cell Lymphoma (MCL), including 20 cases Relapsed/Refractory (R/R) to Bruton Tyrosine kinase inhibitors (BTKi)
Functional study of the B-Cell Receptor (BCR) activity by flow cytometry in Mantle Cell Lymphoma (MCL) cell samples | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Performed on formalin-fixed paraffin-embedded (FFPE) tissue sections as well as, when available, on frozen material or viable cryopreserved cells at Mantle Cell Lymphoma (MCL) diagnosis. The aim is to perform a functional study of the B-Cell Receptor (BCR) activity: multiplexed phospho-specific flow cytometry on 10-20 Relapsed/Refractory (R/R) Mantle Cell Lymphoma cases.
To understand the mechanisms of evasion from B-Cell Receptor (BCR) requirement, with particular focus on Mantle Cell Lymphoma (MCL) cases that are resistant to Chemo-immunotherapy (CIT) and/or Bruton Tyrosine kinase (BTK) inhibition | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Performed on formalin-fixed paraffin-embedded (FFPE) tissue sections as well as, when available, on frozen material or viable cryopreserved cells at Mantle Cell Lymphoma (MCL) diagnosis. The aim is to understand the mechanisms of evasion from B-Cell Receptor (BCR) requirement as follow:
  * Immunoglobulin (IgH/IgL V(D)J) profiling by Next Generation Sequencing (NGS) on 80 mantle cell lymphoma (MCL) cases;
  * Chromatin accessibility studies (Assay for Transposase-Accessible Chromatin sequencing, ATAC-seq) on approximately 20 cases among the Immunoglobulin (Ig)-negative identified cases or Bruton Tyrosine kinase inhibitors (BTKi) refractory cases, irrespective of their B-Cell Receptor (BCR) status, and on other 20 cases, from the group of patients sensitive to Bruton Tyrosine kinase inhibitors (BTKi);
  * Gene Expression Profiling (GEP) by RNA-seq, on about 20 cases selected on the basis of results of the Assay for Transposase-Accessible Chromatin sequencing (ATAC-Seq) analysis;
Unveil the role of the MALT1-MYC (Mucosa-associated lymphoid tissue lymphoma translocation protein 1 - MYC) pathway in Mantle Cell Lymphoma (MCL) cases expressing or not the BCR (B-Cell Receptor) | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Performed on formalin-fixed paraffin-embedded (FFPE) tissue sections as well as, when available, on frozen material or viable cryopreserved cells at Mantle Cell Lymphoma (MCL) diagnosis. The aim is to perform RNA studies on 20 cases
To correlate results of biologic studies with clinical characteristics of patients | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  About 80 cases of Relapsed/Refractory (R/R) Mantle Cell Lymphoma (MCL) with available tissue samples will be considered for correlation between biological studies with clinical characteristics of patients, response to treatment and conventional outcomes (Progression Free Survival, Progression Free Survival at 2 years, Overall Survival, Overall Survival at 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Maria Quaglia, Principal Investigator — Azienda Ospedaliera Universitaria (AOU) Integrata di Verona - Unità Operativa di Ematologia
Locations (16):
- Italy (16):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - AOU Senese - U.O.C. Ematologia, Siena, SI
  - Centro Riferimento Oncologico - S.O.C. Oncologia Medica A, Aviano
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - A.O. S. Croce e Carle, Cuneo
  - Azienda Ospedaliera Universitaria Careggi- Unità funzionale di ematologia, Florence
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - AOU di Padova - Ematologia, Padua
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia - Ematologia, Reggio Emilia
  - A.O.U. Citta della Salute e della Scienza di Torino- Ematologia Universitaria, Torino
  - Ospedale Ca' Foncello - S.C di Ematologia, Treviso
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ematologica, Udine
  - AOU Integrata di Verona - U.O. Ematologia, Verona
  - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided